CLINICAL TRIAL: NCT02538549
Title: A Pilot Randomized Controlled Trial to Test Effectiveness of the ACE4 (Activity Challenge - 4 Areas) for Depression and Anxiety: A Behavioural Activation Based Game.
Brief Title: Pilot RCT to Test Effectiveness of the ACE4 (Activity Challenge- 4 Areas) for Depression and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Farooq Naeem, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 6015291
Record Dates: First submitted 2015-08-29; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Anxiety Disorder; Mixed With Depression (Mild)
MeSH Terms: conditions — Anxiety Disorders; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACE4 and TAU (Active Comparator): This group will receive ACE4 as an intervention and treatment as usual.
  Interventions: Behavioral: ACE4
- TAU Only (No Intervention): This group will receive only the treatment as usual.

INTERVENTIONS:
Behavioral: ACE4 — Activity Challenge 4 is a single player card game that is based on principles of behavioral activation. The game was used with crisis and transitional case management clients, with positive feedback.
  Arms: ACE4 and TAU

SUMMARY:
Behavioral activation (BA) is a low cost, evidence-based intervention that can be effective in treating depression and anxiety. We have developed a behavioural activation card game for clients receiving treatment through the Crisis Team and Traditional Case Management (TCM) in Kingston, ON. The game is designed to integrate behavioural activation tools into daily life while receiving points for completion of the each Activity Challenge, which are divided into 4 areas (ACE4), with the goal to receive maximum amount of points in the timeframe of the study. Using a Randomized Control Trial (RCT) design, participants (n=40) will be assigned to one of two groups, with the intervention group receiving ACE4 and treatment as usual (TAU) and the control group only receiving TAU. Assessments will be carried out upon entry to the study and at the end of the intervention period (8 weeks). Assessments will be completed using the WHODAS 2.0 (World Health Organization Disability Assessment Schedule), HADS (The Hospital Anxiety and Depression Scale), and CORE (Clinical Outcome in Routine Evaluation). We hypothesize that the treatment group receiving the ACE4 intervention will show improvement in overall mental state. Analyses will be conducted using SPSSv16, an analysis of covariance and t-test, and a binary logistic regression analysis will be used to investigate factors that predict good outcomes. Results will be published in international journals and presented at conferences with an aim towards being applied to clinics in Pakistan.

DETAILED DESCRIPTION:
INTRODUCTION:

Behavioral activation (BA) is an evidence based intervention that has been found to be effective in treating depression (ref). It has the advantage of being low cost and can be used by people with low literacy. BA can be easily delivered in low and middle income countries like Pakistan, if appropriately adapted.

We have developed a single player card game that is based on principles of behavioral activation. The game was used with crisis and transitional case management clients, with positive feedback. This is a pilot study using a RCT design to test the effectiveness of this game.

Objective To assess effectiveness of ACE4, for depression against care as usual. Study design and duration This study is a Randomized Controlled Trial (RCT) which aims to assess effectiveness of ACE4 against care as usual for depression. Study participants will be randomly assigned to two groups the intervention group will receive ACE4 and TAU, while the control group will receive only TAU.

ACE4: Introduction Intervention focuses on behavioral activation. Although ACE4 is a single player game, it can be facilitated by a carer. The game comes with 15 cards in four colour, with each colour representative of an activity area (for example, Creative activities, recreational, self care and work, social and spiritual activities). The idea is to choose equal number of activities from each colour. Every card has a number. Patients have to write this number on activity calendar that comes with this game, along with the time activity was performed. The aim of the game is to score maximum points at the end of the 6 weeks. Those with scores in high range get ACE4 badge (in addition to getting an improvement in their mood)

Inclusion and exclusion criteria All those who fulfill the diagnostic criteria of Depressive episode (F32) or Recurrent depressive disorder (F33 except 33.4 ) using ICD10 RDC (based on interviews using SCAN Urdu version), are between the ages of 18 to 65, score 8 or more on HADS, Depression Subscale, will be approached. Patients will be asked to attend a further appointment at the end of study period and will be assessed again.

The exclusion criteria include; excessive use of alcohol or drugs (using ICD 10 RDC for alcohol or drug abuse or dependence) significant cognitive impairment (for example learning disability or dementia) and active psychosis.

Procedure Patients who have been referred for the study will be provided brief information about the study. Those who meet the criteria and consent will be then asked to join the study and will be allocated to one arm of the trial after randomization.

Sample size This is a feasibility study. We will take 40 patients, with 20 in each arm.

Randomization Randomization will be performed distantly by a statistician, from the list of all the patients who have been accepted for each group. After randomization patients will be allocated to either treatment or the control arm. Randomization will be performed for each group separately.

INSTRUMENTS The assessments will be carried out at the base line and then at the end of therapy (8 weeks). Control group will receive care as usual.A number equal to intervention group will be employed in this group. Blind raters will be used to assess the change in depression.

The Hospital Anxiety and Depression Scale (HAD) (Zigmond and Snaith, 1983) is a 14 item, self assessment scale designed to measure anxiety and depression. It has a high internal consistency, face validity and concurrent validity. Even-numbered questions relate to depression and odd-numbered questions relate to anxiety. Each question has 4 possible responses. Responses are scored on a scale from 3 to 0. The maximum score is therefore 21 for depression and 21 for anxiety. A score of 11 or higher indicates the probable presence of the mood disorder with a score of 8 to 10 being just suggestive of the presence of the respective state. The two subscales, anxiety and depression, have been found to be independent measures. In its current form the HADS is now divided into four ranges: normal (0-7), mild (8-10), moderate (11-15) and severe (16-21).

The Clinical Outcome in Routine Evaluatoin (CORE) is is a client self-report questionnaire designed to be administered before and after therapy. The client is asked to respond to 34 questions about how they have been feeling over the last week, using a 5-point scale ranging from 'not at all' to 'most or all of the time'. The 34 items of the measure cover four dimensions: Subjective well-being, Problems/symptoms, Life functioning and Risk/harm. The responses are designed to be averaged by the practitioner to produce a mean score to indicate the level of current psychological global distress (from 'healthy' to 'severe'). The questionnaire is repeated after the last session of treatment; comparison of the pre-and post-therapy scores offers a measure of 'outcome' (i.e. whether or not the client's level of distress has changed, and by how much) (Evans, 2000).

Brief Disability Questionnaire (BDQ) was developed by the WHO to measure disability due to physical and psychological problems and has been used extensively in research (Von Korff et al., 1996).

A data form will be used to collect information from the client.

Study sites Crisis and the TCM services in Kingston, ON, Canada.

Data entry and analysis Statistical analyses would be carried out using an intention to treat. Analyses will be carried out using SPSS v16 . Both parametric and non parametric tests will be carried out as appropriate to compare groups. An analysis of covariance will be used to measure the differences between the two groups at three time points, where the data is normally distributed. A t test will be used to compare groups, both paired and un-paired. SPSS frequency and descriptive commands will be used to measure descriptive statistics. SPSS explore command will be used to measure normality of the data, using histograms and Kolmorogov Smirnov test. If the therapy is proved to be more effective than the control, we will also use a binary logistic regression analysis to explore factors which predict good outcome. An intention to treat analysis will be performed. Number Needed to Treat (NNT) will be calculated to assist clinicians with clinical decision making.

Research in clinically naturalistic settings It is recognized that such research is most likely to provide results that are relevant to routine clinical practice; the current study provides a more rigorous evaluation for an intervention that can be provided in current service in Pakistan and at no extra costs.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the diagnostic criteria of Depressive episode (F32) or Recurrent depressive disorder (F33 except 33.4 ) using ICD10 RDC (based on interviews using SCAN Urdu version).
* Between the ages of 18 to 65
* Score 8 or more on HADS, Depression Subscale.
* Patients will be asked to attend a further appointment at the end of study period and will be assessed again.

Exclusion Criteria:

* Excessive use of alcohol or drugs (using ICD 10 RDC for alcohol or drug abuse or dependence).
* Significant cognitive impairment (for example learning disability or dementia).
* Active psychosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The Hospital Anxiety and Depression Scale (HAD) | At the base line and then at the end of therapy (8 weeks).
  A 14 item, self assessment scale designed to measure anxiety and depression. It has a high internal consistency, face validity and concurrent validity. Even-numbered questions relate to depression and odd-numbered questions relate to anxiety. Each question has 4 possible responses. Responses are scored on a scale from 3 to 0. The maximum score is therefore 21 for depression and 21 for anxiety. A score of 11 or higher indicates the probable presence of the mood disorder with a score of 8 to 10 being just suggestive of the presence of the respective state. The two subscales, anxiety and depression, have been found to be independent measures. In its current form the HADS is now divided into four ranges: normal (0-7), mild (8-10), moderate (11-15) and severe (16-21).

SECONDARY OUTCOMES:
The Clinical Outcome in Routine Evaluation (CORE) | At the base line and then at the end of therapy (8 weeks).
  a client self-report questionnaire designed to be administered before and after therapy. The client is asked to respond to 34 questions about how they have been feeling over the last week, using a 5-point scale ranging from 'not at all' to 'most or all of the time'. The 34 items of the measure cover four dimensions: Subjective well-being, Problems/symptoms, Life functioning and Risk/harm. The responses are designed to be averaged by the practitioner to produce a mean score to indicate the level of current psychological global distress (from 'healthy' to 'severe'). The questionnaire is repeated after the last session of treatment; comparison of the pre-and post-therapy scores offers a measure of 'outcome' (i.e. whether or not the client's level of distress has changed, and by how much).
Brief Disability Questionnaire (BDQ) | At the base line and then at the end of therapy (8 weeks).
  Developed by the WHO to measure disability due to physical and psychological problems and has been used extensively in research.

CONTACTS AND LOCATIONS:
Overall Officials: Farooq Naeem, MsC, PhD, Principal Investigator — Queen's University
Locations (1):
- Addiction & Mental Health Services - Kingston Frontenac Lennox & Addington, Kingston, Ontario, Canada